CLINICAL TRIAL: NCT01139411
Title: Parental Involvement as a Strategy to Enhance Adolescent Weight Control
Brief Title: The Role of Parents in Adolescent Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Elissa Jelalian, Senior Scientist, The Miriam Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GRANT00538804; R03HD060137 (NIH)
Record Dates: First submitted 2010-06-07; First posted 2010-06-08 (Estimated); Results first posted 2016-09-30 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-08

CONDITIONS: Adolescent Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Behavioral Weight Control with Enhanced Parent Involvement (Experimental): This treatment arm included periodic dyadic sessions with adolescents and their parents, focusing on weight-related communication combined with standard behavioral weight control.
  Interventions: Behavioral: Behavioral Weight Control with Enhanced Parent Involvement
- Behavioral Weight Control with Minimal Parent Involvement (Placebo Comparator): This treatment arm included standard behavioral weight control delivered to the adolescent with minimal parent involvement.
  Interventions: Behavioral: Behavioral Weight Control with Minimal Parent Involvement

INTERVENTIONS:
Behavioral: Behavioral Weight Control with Enhanced Parent Involvement
  Arms: Behavioral Weight Control with Enhanced Parent Involvement
Behavioral: Behavioral Weight Control with Minimal Parent Involvement
  Arms: Behavioral Weight Control with Minimal Parent Involvement

SUMMARY:
The purpose of the study is to determine whether a novel model of including parents in adolescent weight control results in greater decrease in adolescent z-BMI compared to an intervention with minimal parent involvement.

ELIGIBILITY:
Inclusion Criteria:

* Between 30 and 90% overweight
* Parent or guardian willing to participate

Exclusion Criteria:

* Major psychiatric disorder

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 49 (Actual)
Dates: Start 2009-08; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Miriam Hospital, Providence, Rhode Island, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Behavioral Weight Control With Minimal Parent Involvement: This treatment arm included standard behavioral weight control delivered to the adolescent with minimal parent involvement.
  Behavioral Weight Control with Minimal Parent Involvement
- Behavioral Weight Control With Enhanced Parent Involvement: This treatment arm included periodic dyadic sessions with adolescents and their parents, focusing on weight-related communication combined with standard behavioral weight control.
  Behavioral Weight Control with Enhanced Parent Involvement
Period: Overall Study
Arm/Group | Behavioral Weight Control With Minimal Parent Involvement | Behavioral Weight Control With Enhanced Parent Involvement
Started | 26 | 23
Completed | 24 | 19
Not Completed | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Behavioral Weight Control With Enhanced Parent Involvement | Behavioral Weight Control With Minimal Parent Involvement | Total
Number analyzed (Participants) | 23 | 26 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 23 | 26 | 49
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.21 (1.40) | 15.00 (1.30) | 15.10 (1.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 17 | 37
  Male | 3 | 9 | 12
Region of Enrollment [Number; unit: participants]
  United States | 23 | 26 | 49
Body Mass Index (kg/m^2) [Mean (Standard Deviation); unit: kilograms/meters squared (kg/m2)] | 33.25 (4.02) | 31.17 (3.01) | 32.16 (3.64)
Parent modeling 1: Dietary Choices (WCSS) [Mean (Standard Deviation); unit: units on a scale] — Parent modeling of dietary choices was assessed using the Diet Choices subscale of the Weight Control Strategies Scale (WCSS), a parent-report measure of his/her own healthy weight control practices. The Dietary choices subscale of the WCSS has a scale range of 0 - 4, with higher scores corresponding to healthier diet choices.
  units on a scale | 2.70 (0.76) | 2.32 (1.13) | 2.50 (0.98)
Parent modeling 2: Self-monitoring (WCSS) [Mean (Standard Deviation); unit: units on a scale] — Parent modeling of self-monitoring behavior was assessed using the Self Monitoring subscale of the Weight Control Strategies Scale (WCSS), a parent-report measure of his/her own healthy weight control practices. The Self Monitoring subscale of the WCSS has a scale range of 0 - 4, with higher scores corresponding to more self-monitoring behavior.
  units on a scale | .81 (0.80) | 0.55 (0.70) | 0.67 (0.75)
Parent modeling 3: Physical Activity (WCSS) [Mean (Standard Deviation); unit: units on a scale] — ). Parent modeling of Physical Activity was assessed using the Physical Activity subscale of the Weight Control Strategies Scale (WCSS), a parent-report measure of his/her own healthy weight control practices. The Physical Activity subscale of the WCSS has a scale range of 0-4, with higher scores corresponding to greater physical activity.
  units on a scale | 1.75 (1.17) | 0.90 (1.05) | 1.30 (1.18)
Parent modeling 4: Weight and Body Concerns [Mean (Standard Deviation); unit: units on a scale] — Parent modeling of concern about weight/body was assessed using the Parent Modeling of Weight and Body Concerns subscale of the Family Experiences Related to Food Questionnaire (FERF-Q)), an adolescent-report measure of parent behavior pertaining to weight control. The Weight and Body Concerns subscale of the FERF-Q has a scale range of 1 - 5, with greater scores corresponding to greater parent weight and body concerns, as perceived and reported by the adolescent.
  units on a scale | 2.75 (0.80) | 2.90 (0.89) | 2.83 (0.84)
Communication 1: Negative weight-related comments [Mean (Standard Deviation); unit: units on a scale] — Negative maternal weight-related commentary was assessed using the Negative maternal weight-related commentary subscale of the Family Experiences Related to Food Questionnaire (FERF-Q)), an adolescent-report measure of parent behavior pertaining to weight control. The Negative maternal weight-related commentary subscale of the FERF-Q has a scale range of 1 - 5, with higher scores corresponding to greater negative maternal weight-related commentary, as perceived and reported by the adolescent.
  units on a scale | 2.73 (0.73) | 2.85 (0.64) | 2.79 (0.70)
Communication 2: Observed parent-adolescent communication quality [Mean (Standard Deviation); unit: units on a scale] — Observed parent-adolescent communication quality was measured using the Dyadic Observed Communication Scale (DOCS) used to code communication between adolescent and caregiver during a video-taped observational coding session. The DOCS is coded on a scale of 0 -10, with higher scores reflecting higher quality of communication, as observed by an independent rater.
  units on a scale | 5.5 (2.1) | 5.8 (1.9) | 5.7 (1.9)

OUTCOME MEASURES:

1. Primary Outcome: Body Mass Index
Description: Post-treatment BMI (controlling for baseline BMI)
Time Frame: Baseline and at completion of 16 week intervention
Measure: Mean (Standard Deviation); unit: kilograms/meters squared
Arm/Group | Behavioral Weight Control With Minimal Parent Involvement | Behavioral Weight Control With Enhanced Parent Involvement
Number analyzed (Participants) | 26 | 23
kilograms/meters squared | 29.89 (3.41) | 32.82 (4.06)
Statistical Analysis 1: Comparison: Behavioral Weight Control With Minimal Parent Involvement vs Behavioral Weight Control With Enhanced Parent Involvement; Null hypothesis was that the amount of weight lost by adolescents in Enhanced Parent Involvement and Minimal Parent involvement would not be significantly different. The study was powered at .8 to achieve a medium effect size (f = .26; partial eta sq. = 0.06). The end-of-treatment BMI value was the dependent variable, with the baseline BMI value entered as a covariate; Test type: Superiority or Other; p = 0.06, ANCOVA — Threshold for significance: 0.05

2. Secondary Outcome: Parent Modeling 1: Dietary Choices (WCSS)
Description: Post-treatment value (controlling for baseline). Parent modeling of dietary choices was assessed using the Diet Choices subscale of the Weight Control Strategies Scale (WCSS), a parent-report measure of his/her own healthy weight control practices. The Dietary choices subscale of the WCSS has a scale range of 0 - 4, with higher scores corresponding to healthier diet choices. Higher scores are considered to be a better treatment outcome.
Time Frame: Baseline to post-treatment
Population: Secondary outcomes analyzed for treatment completers only.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Behavioral Weight Control With Enhanced Parent Involvement | Behavioral Weight Control With Minimal Parent Involvement
Number analyzed (Participants) | 19 | 24
units on a scale | 2.92 (0.82) | 2.87 (0.50)
Statistical Analysis 1: Comparison: Behavioral Weight Control With Enhanced Parent Involvement vs Behavioral Weight Control With Minimal Parent Involvement; The end-of-treatment value was the dependent variable, with the baseline value entered as a covariate; Test type: Superiority or Other; p = 0.58, ANCOVA — Threshold for significance: 0.05

3. Secondary Outcome: Parent Modeling 2: Self-monitoring (WCSS)
Description: Post-treatment value (controlling for baseline). Parent modeling of self-monitoring behavior was assessed using the Self Monitoring subscale of the Weight Control Strategies Scale (WCSS), a parent-report measure of his/her own healthy weight control practices. The Self Monitoring subscale of the WCSS has a scale range of 0 - 4, with higher scores corresponding to more self-monitoring behavior. Higher scores are thought to reflect a better treatment outcome.
Time Frame: Baseline to post-treatment
Population: Secondary outcomes analyzed for treatment completers only.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Behavioral Weight Control With Minimal Parent Involvement | Behavioral Weight Control With Enhanced Parent Involvement
Number analyzed (Participants) | 24 | 19
units on a scale | 0.81 (0.81) | 1.28 (0.67)
Statistical Analysis 1: Comparison: Behavioral Weight Control With Minimal Parent Involvement vs Behavioral Weight Control With Enhanced Parent Involvement; Test type: Superiority or Other; p = 0.19, ANCOVA — Threshold for significance: 0.05

4. Secondary Outcome: Parent Modeling 3: Physical Activity (WCSS)
Description: Post-treatment value (controlling for baseline). Parent modeling of Physical Activity was assessed using the Physical Activity subscale of the Weight Control Strategies Scale (WCSS), a parent-report measure of his/her own healthy weight control practices. The Physical Activity subscale of the WCSS has a scale range of 0-4, with higher scores corresponding to greater physical activity. Higher scores are considered a better treatment outcome.
Time Frame: Baseline to post-treatment
Population: Secondary outcomes analyzed for treatment completers only
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Behavioral Weight Control With Enhanced Parent Involvement | Behavioral Weight Control With Minimal Parent Involvement
Number analyzed (Participants) | 19 | 24
units on a scale | 1.9 (1.0) | 1.32 (0.75)
Statistical Analysis 1: Comparison: Behavioral Weight Control With Enhanced Parent Involvement vs Behavioral Weight Control With Minimal Parent Involvement; Test type: Superiority or Other; p = 0.72, ANCOVA — Threshold for significance: 0.05

5. Secondary Outcome: Parent Modeling 4: Weight and Body Concerns (FERF-Q)
Description: Post-treatment value (controlling for baseline). Parent modeling of concern about weight/body was assessed using the Parent Modeling of Weight and Body Concerns subscale of the Family Experiences Related to Food Questionnaire (FERF-Q)), an adolescent-report measure of parent behavior pertaining to weight control. The Weight and Body Concerns subscale of the FERF-Q has a scale range of 1 - 5, with higher scores corresponding to greater parent weight and body concerns, as perceived and reported by the adolescent. Lower weight and body concern is considered a better treatment outcome.
Time Frame: Baseline to post-treatment
Population: Secondary outcomes analyzed for treatment completers only
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Behavioral Weight Control With Enhanced Parent Involvement | Behavioral Weight Control With Minimal Parent Involvement
Number analyzed (Participants) | 19 | 24
units on a scale | 2.63 (1.02) | 2.64 (0.88)
Statistical Analysis 1: Comparison: Behavioral Weight Control With Enhanced Parent Involvement vs Behavioral Weight Control With Minimal Parent Involvement; Test type: Superiority or Other; p = 0.41, ANCOVA

6. Secondary Outcome: Communication 1: Negative Maternal Weight-related Commentary (FERF-Q)
Description: Post-treatment value (controlling for baseline). Negative maternal weight-related commentary was assessed using the Negative maternal weight-related commentary subscale of the Family Experiences Related to Food Questionnaire (FERF-Q)), an adolescent-report measure of parent behavior pertaining to weight control. The Negative maternal weight-related commentary subscale of the FERF-Q has a scale range of 1 - 5, with higher scores corresponding to greater negative maternal weight-related commentary, as perceived and reported by the adolescent. Lower scores are considered a better treatment outcome.
Time Frame: Baseline to post-treatment
Population: Secondary outcomes analyzed for treatment completers only
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Behavioral Weight Control With Enhanced Parent Involvement | Behavioral Weight Control With Minimal Parent Involvement
Number analyzed (Participants) | 19 | 24
units on a scale | 2.71 (0.80) | 2.32 (0.70)
Statistical Analysis 1: Comparison: Behavioral Weight Control With Enhanced Parent Involvement vs Behavioral Weight Control With Minimal Parent Involvement; Test type: Superiority or Other; p = 0.01, ANCOVA — Threshold for significance: 0.05

7. Secondary Outcome: Communication 2: Observed Parent-adolescent Communication Quality (DOCS)
Description: Post-treatment value (controlling for baseline). Observed parent-adolescent communication quality was measured using the Dyadic Observed Communication Scale (DOCS) used to code communication between adolescent and caregiver during a video-taped observational coding session. The DOCS is coded on a scale of 0 -10, with higher scores reflecting higher quality of communication, as observed by an independent rater. Higher scores are thought to reflect a better treatment outcome.
Time Frame: Baseline to post-treatment
Population: 38 participants (19 in each group) had complete baseline and post treatment data for videotaped observations.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Behavioral Weight Control With Enhanced Parent Involvement | Behavioral Weight Control With Minimal Parent Involvement
Number analyzed (Participants) | 19 | 19
units on a scale | 5.5 (1.9) | 5.8 (1.8)
Statistical Analysis 1: Comparison: Behavioral Weight Control With Enhanced Parent Involvement vs Behavioral Weight Control With Minimal Parent Involvement; Test type: Superiority or Other; p = 0.61, ANCOVA — Threshold for significance: 0.05

ADVERSE EVENTS:
Time Frame: Baseline through post-treatment (4 months)
Arm/Group | Behavioral Weight Control With Minimal Parent Involvement | Behavioral Weight Control With Enhanced Parent Involvement
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/23
Other Adverse Events (participants affected / at risk) | 0/26 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No